CLINICAL TRIAL: NCT04282590
Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of TRK-750 in Colorectal Cancer Patients With Chemotherapy-induced Peripheral Neuropathy Following Oxaliplatin-containing Chemotherapy in the Adjuvant Setting
Brief Title: A Study to Investigate the Safety and Efficacy of TRK-750 for the Treatment of Patients With CIPN (Chopin Study)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: due to COVID-19 pandemic
Sponsor: Toray Industries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 750CNP01
Record Dates: First submitted 2020-02-17; First posted 2020-02-25 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Period 1: TRK-750, Treatment Period 2: placebo (Experimental)
  Interventions: Drug: TRK-750/Placebo
- Treatment Period 1: placebo, Treatment Period 2: TRK-750 (Experimental)
  Interventions: Drug: Placebo/TRK-750

INTERVENTIONS:
Drug: TRK-750/Placebo — Powder for oral solution
  Arms: Treatment Period 1: TRK-750, Treatment Period 2: placebo
Drug: Placebo/TRK-750 — Powder for oral solution
  Arms: Treatment Period 1: placebo, Treatment Period 2: TRK-750

SUMMARY:
The primary objective of the study is:

• to assess the safety and tolerability of multiple oral (twice daily [BID]) doses of TRK-750 in oxaliplatin-treated colorectal cancer patients with chemotherapy-induced peripheral neuropathy (CIPN).

The secondary objectives of the study are:

* to assess the efficacy of multiple oral (BID) doses of TRK-750 in reducing neuropathic symptoms, improving quality of life (QoL), and clinician-reported outcomes in oxaliplatin-treated colorectal cancer patients with CIPN.
* to study the relationship between plasma concentrations of TRK-750 and safety and efficacy variables in oxaliplatin-treated colorectal cancer patients with CIPN.

The exploratory objective of this study is:

• to assess the efficacy of multiple oral (BID) doses of TRK-750 on pharmacodynamic (PD) biomarker(s) in blood, psychophysical, electrophysiological, and histological parameters of neuropathy in oxaliplatin-treated colorectal cancer patients with CIPN.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient between 18 and 80 years of age, inclusive.
2. Oxaliplatin-containing chemotherapy treatment for colorectal cancer in the adjuvant setting must have been completed ≥ 3 months, but not more than 3 years, prior to Screening.
3. A diagnosis of CIPN based on the following criteria:

   1. onset of pain of any severity in hands and/or feet after exposure to oxaliplatin AND;
   2. presence of painful symptoms of any severity in a symmetrical stocking and glove distribution beginning in lower extremities, which may progress to the upper extremities (the latter may or may not be present at study entry) AND;
   3. painful symptoms are accompanied by non-painful symptoms (e.g., tingling or numbness) in a similar distribution.
4. Neuropathy of ≥ Grade 2 using the general guideline of grading scales defined in CTCAE (v5.0)
5. Pain or neuropathic symptoms of CIPN for a duration of ≥ 3 months, for which the patient wants intervention.
6. Body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive.
7. Females of childbearing potential will agree to use highly effective contraception (Appendix 4) from the time of signing the ICF until 90 days after the Follow-up visit. Males who are sexually active with female partners of childbearing potential will agree to use a male condom with spermicide from Day 1 until 90 days after the Follow-up visit.
8. Be either CIPN pain-treatment naïve or have important side effects or inadequate relief from their current CIPN pain medication (stable over last month).
9. Has not used non-pharmacological therapy for the treatment of any pain condition (e.g., chiropractic therapies, alternative medicine therapies, or acupuncture) for at least 2 weeks prior to start of the baseline days (Days -14 to -1), and a willingness to refrain from using these therapies throughout the study. The use of physical activity or other short-acting, symptomatic non-pharmacological therapy is permitted provided the patient is willing to maintain the same regimen or usage pattern consistently throughout the study.
10. Able to comprehend and willing to sign an Informed Consent Form (ICF) and to abide by the study restrictions.
11. Patients have a life expectancy of at least 12 months.
12. An EORTC QLQ-CIPN20 score of ≥ 25 based on an average of 2 assessments during the Screening period and Day 1 prior to randomisation.
13. At least one of the following:

    1. a mean value of pain intensity ≥ 4 on the 11-point NRS based on the average of once-daily assessments for 7 days, with no more than 2 missing records, between Days -7 and -1. Patients must score ≥ 4 on at least 4 out of 7 measurements between Days -7 and -1 OR;
    2. a mean value of intensity of tingling and numbness or uncomfortable neuropathic symptoms ≥ 4 on the 11-point NRS based on the average of once-daily assessments for 7 days, with no more than 2 missing records, between Days -7 and -1. Patients must score ≥ 4 on at least 4 out of 7 measurements between Days -7 and -1.

Exclusion Criteria:

1. Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol, ability to complete the study, and study assessments.
2. Presence of skin conditions in the affected dermatome that, in the judgement of the Investigator, could interfere with evaluation of the neuropathic pain condition.
3. Presence of non-CIPN pain that may interfere with study assessments and/or self-evaluation of peripheral neuropathic pain.
4. Known history of significant hypersensitivity, intolerance, or allergy.
5. Peripheral neuropathy caused by tumour infiltration or compression of spinal nerves or surgical trauma.
6. Active clinically significant infection
7. Unstable cardiac disease or myocardial infarction within 6 months prior to study entry.
8. Patients with uncontrolled major psychiatric disorders, such as major depression or psychosis.
9. History of pre-existing symptomatic neuropathy prior to chemotherapy, including neuropathy due to alcoholism, vitamin B deficiency, diabetes, hypothyroidism, human immunodeficiency virus (HIV), congenital neuropathy, and toxic neuropathy.
10. Female patients who are pregnant (including a positive urine pregnancy test at Screening or on Day 1) or lactating.
11. Inadequate haematological function, defined as neutrophil count < 1.0 × 10^9/L and platelet count < 50 × 10^9/L with measured values of these in the clinical laboratory tests conducted at Screening. At Screening, haematology assessments may be repeated once.
12. Inadequate renal function, defined as estimated glomerular filtration rate (eGFR) ≤ 59 mL/min, i.e., Creatinine Clearance (CrCl) as calculated using the Cockcroft-Gault equation with measured values of these in the clinical laboratory tests conducted at Screening:

    1. [1.23 × (140 - age) × (weight in kg)] ÷ (serum creatinine in μmol/L) - if male.
    2. [1.04 × (140 - age) × (weight in kg)] ÷ (serum creatinine in μmol/L) - if female.

    At Screening, clinical laboratory assessments may be repeated once.
13. History of alcoholism or drug/chemical abuse within 1 year prior to Day 1.
14. Positive test results for drugs of abuse at Screening (confirmed by repeat) or Day 1, unless consistent with use of prescription medication and approved by the Sponsor (or delegate). A repeated positive test result for cocaine, phencyclidine, methadone, or amphetamines, for nonmedical use, are unconditionally exclusionary.
15. Positive test for hepatitis B surface antigen (HbsAg), hepatitis C antibody (HCV), or HIV antibody at Screening.
16. Use of any medication in the absence of appropriate washout periods that, in the opinion of the Investigator, may influence the result of the study, or the patient's ability to participate in the study.
17. Has received an investigational product or has been treated with an investigational device within 90 days prior to first drug administration and will not start any other investigational product or device study within 90 days after last study drug administration.
18. Likely to require chemotherapy during the study period or any other treatment that may interfere with compliance with the protocol, ability to complete the study, and study assessments.
19. Plans to change current medications or any other intervention intended to treat or relieve CIPN signs or symptoms from Screening to end of study.
20. Has previously received TRK-750.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events as assessed by CTCAE v5.0 | Up to Week 28
Proportion of patients with clinically significant changes in vital signs: supine blood pressure (mmHg), supine pulse rate (beats/min), respiratory rate (breaths/min), and oral body temperature (°C or °F) | Up to Week 28
Proportion of patients with clinically significant changes in electrocardiogram time intervals | Up to Week 24
Proportion of patients with clinically significant changes in clinical laboratory tests | Up to Week 28

SECONDARY OUTCOMES:
Absolute change and percentage change of Numerical Rating Scale (NRS) from baseline in neuropathic symptoms | Week 12
  Pain and distressing neuropathic symptoms intensities will be assessed for neuropathic symptoms.
  * for pain intensity: weekly average of NRS daily (evening) assessments.
  * for distressing neuropathic symptoms such as tingling and numbness intensity: weekly average of NRS of daily (evening) assessments.
Proportion of patients with a reduction of at least 30% relative to baseline in neuropathic symptoms intensity on weekly average of NRS daily assessments | Week 12
Change from baseline in EORTC QLQ-CIPN20 patient-reported outcome scale | Week 12
Proportion of patients with 2 points or more improvement relative to baseline in EORTC QLQ-CIPN20 sensory subscale assessments | Week 12
Change from baseline in EORTC QLQ-C30 | Week 12
Change from baseline in TNSc | Week 12
Change from baseline in CTCAE (v5.0) neuropathy grade. | Week 12
Plasma concentrations of TRK-750 (ng/mL) | Up to Week 28

OTHER OUTCOMES:
Change from baseline in QST parameter: cold detection threshold (°C) | Week 12
  The assessment will be study site dependent. For sites with the ability to perform the assessment, all patients will be evaluated.
Change from baseline in QST parameter: warm detection threshold (°C) | Week 12
  The assessment will be study site dependent. For sites with the ability to perform the assessment, all patients will be evaluated.
Change from baseline in QST parameter: mechanical detection threshold (Von Frey filament detection [g]) | Week 12
  The assessment will be study site dependent. For sites with the ability to perform the assessment, all patients will be evaluated.
Change from baseline in QST parameter: vibration disappearance threshold (Hz) | Week 12
  The assessment will be study site dependent. For sites with the ability to perform the assessment, all patients will be evaluated.
Change from baseline in QST parameter: cold pain threshold (°C) | Week 12
  The assessment will be study site dependent. For sites with the ability to perform the assessment, all patients will be evaluated.
Change from baseline in QST parameter: heat pain threshold (°C) | Week 12
  The assessment will be study site dependent. For sites with the ability to perform the assessment, all patients will be evaluated.
Change from baseline in QST parameter: mechanical pain threshold (mN) | Week 12
  The assessment will be study site dependent. For sites with the ability to perform the assessment, all patients will be evaluated.
Change from baseline in QST parameter: pressure pain threshold (kPa) | Week 12
  The assessment will be study site dependent. For sites with the ability to perform the assessment, all patients will be evaluated.
Change from baseline in electrophysiological amplitude in the sural, superficial radial, and tibial nerves: motor nerve (mV) | Week 12
  The assessment will be study site dependent. For sites with the ability to perform the assessment, all patients will be evaluated.
Change from baseline in electrophysiological amplitude in the sural, superficial radial, and tibial nerves: sensory nerve (microV) | Week 12
  The assessment will be study site dependent. For sites with the ability to perform the assessment, all patients will be evaluated.
Change from baseline in electrophysiological conduction velocity (m/sec) in the sural, superficial radial, and tibial nerves | Week 12
  The assessment will be study site dependent. For sites with the ability to perform the assessment, all patients will be evaluated.
Restoring nerve fiber phenotype in punch skin biopsies (mm) | Week 12
  The assessment will solely be at the discretion of the patient.
Change from baseline in Neurofilament Light Chain (pg/mL) | Week 12